CLINICAL TRIAL: NCT05057234
Title: PRecision Oncology Evidence Development in Cancer Treatment - Liquid AKA the Real World Clinical Utility of ctDNA Analysis for Decision Making and Access to Precision Therapy for Advanced Cancer Patients in BC: The RAPTor Sub-study
Brief Title: PRecision Oncology Evidence Development in Cancer Treatment - Liquid
Acronym: PREDiCTl
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PREDiCTl
Record Dates: First submitted 2021-07-02; First posted 2021-09-27 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: next generation sequencing panel; cost consequence; liquid biopsy; ctDNA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Simultaneous - FoundationOne liquid CDx (Experimental): Patients undergoing FoundationOne liquid CDx while tissued-based NGS panel is in progress or reported within 4 weeks of enrollment
  Interventions: Diagnostic Test: FoundationOne liquid CDx; Behavioral: Quality of life questionnaires
- Simultaneous - no additional testing (Experimental): Patients undergoing no additional testing while tissue-based NGS panel is in progress or reported within 4 weeks of enrolment
  Interventions: Behavioral: Quality of life questionnaires
- Sequential - FoundationOne liquid CDx (Experimental): Patients undergoing FoundationOne liquid CDx if standard tissue based NGS oncopanel testing identifies no somatic tier 1 variant of strong clinical significance
  Interventions: Diagnostic Test: FoundationOne liquid CDx; Behavioral: Quality of life questionnaires

INTERVENTIONS:
Diagnostic Test: FoundationOne liquid CDx — FoundationOne liquid CDx testing
  Arms: Sequential - FoundationOne liquid CDx; Simultaneous - FoundationOne liquid CDx
Behavioral: Quality of life questionnaires — Quality of life questionnaire - EQ5D

SUMMARY:
The current standard of care for molecular characterization of tumors is tissue based next generation sequencing (NGS) panel. Liquid biopsies (ie blood) are of increasing interest and have been implemented as a diagnostic tool in some countries. This study compares tissue based and liquid based testing to evaluate the detection rate and cost consequence of using this new tool in BC.

DETAILED DESCRIPTION:
Part A - Simultaneous - Patients will be randomized 1:1 to FoundationOne liquid CDx or no additional testing simultaneously at initiation of request for standard based tissue based next generation sequencing (NGS) panel testing. The objective of Part A is to evaluate the cost-consequence of the liquid ctDNA biopsy technology, FoundationOne liquid CDx, for first line molecular characterization of advanced colorectal cancer, melanoma, non small cell lung cancer (NSCLC), ovarian cancer, prostate cancer and triple negative breast cancer with simultaneous molecular characterization by tissue based NGS panel

Part B - Sequential - Patients will undergo standard tissue based NGS panel testing and if there are no somatic tier 1 variant of strong clinical significance identified the patients will then be eligible for FoundationOne liquid CDx. The objective of Part B is to determine the benefit of a sequential approach with molecular characterization by tissue based NGS panel testing followed by liquid based FoundationOne liquid CDx for patients who do not have an actionable tissue based oncogenic driver, across British Columbia.

The development and access to next generation sequencing (NGS) technologies on tumour tissue and blood allows the ability to profile the genomic landscape of the tumour within reasonable turn-around times and costs. The promise of precision oncology is the ability to 'match the right drug to the right patient at the right time'. Despite considerable excitement at the prospect of genome-informed therapy to improve oncologic outcomes, there has been little empirical assessment of its benefit from an overall population perspective and its true impact on cancer care delivery in 'real-world' scenarios.

While the enthusiasm for liquid biopsies has increased, the understanding of the cost implications lags behind. We propose to assess the true clinical impact on both individual patients and on a population-based cancer system of precision oncology via ctDNA analyses in metastatic solid tumors in a real-world scenario.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Patients with metastatic malignancy
* Patients undergoing tissue based molecular characterization by tissue based NGS panel

Part A - Simultaneous

* Tissue based NGS panel requested or reported within 4 weeks of enrolment
* Patients receiving treatment at BC Cancer

Part B - Sequential

* Tissue based NGS oncopanel does NOT identify a somatic tier 1 variant of strong clinical significance OR fails/not feasible due to insufficient tissue
* BC Cancer - Provincial (not including Vancouver Centre)

Exclusion Criteria:

* Patients not available for follow up
* Patients who are not willing to consider systemic treatment options

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Simultaneous: 12-month health resource utilization | 12 months
  To compare health resource utilization of tissue based NGS panel alone, versus NGS panel and FoundationOne liquid CDx measured in Canadian dollars
Sequential: Proportion of patients with an actionable sequencing result following uninformative standard care oncopanel results, treated at BC Cancer, outside Vancouver Centre. | 24 months
  To evaluate the ability of FoundationOne liquid CDx to detect actionable mutations that were not identified on the tissue based NGS oncopanel.

SECONDARY OUTCOMES:
Simultaneous: 18 and 24-month health resource utilization | 24 months
  To evaluate the health resource utilization of tissue based NGS panel alone, versus panel and FoundationOne liquid CDx measured in Canadian dollars
Simultaneous: Clinical utility | 24 months
  To evaluate the clinical utility of tissue based NGS oncopanel +/- FoundationOne liquid CDx as measured by concordance/discordance of findings and subsequent treatment
Simultaneous: Diagnostic pathway impact | 24 months
  To assess the impact of FoundationOne liquid CDx on the diagnostic patient pathway by comparing the number of patients who require repeat biopsies for molecular characterization.
Simultaneous: Quality of Life | 24 months
  To compare the quality of life impact of FoundationOne liquid CDx using the validated instrument, EuroQol 5 Dimension (EQ5D) (Scale of 0-100 where 0 is worst health and 100 is best health)
Sequential: Clinical utility | 24 months
  To evaluate the clinical utility of tissue based NGS oncopanel followed by FoundationOne liquid CDx as measured by concordance/discordance of findings and subsequent treatment
Sequential: Proportion of patients with insufficient tissue for molecular characterization | 24 months
  To determine the proportion of tissue based NGS oncopanel completed for which results are not available due to insufficient tissue. To be calculated by assessing number of patients with insufficient tissue for molecular characterization over the number of patients who have molecular characterization performed

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Ho, MD, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada